CLINICAL TRIAL: NCT04887545
Title: Immune- and Microenvironment- Proteogenomics Profiling for Classifying Lung Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Hospital Cuf Descobertas (Unknown)
Responsible Party: Principal Investigator, Rune Matthiesen, Principal Investigator, Universidade Nova de Lisboa
Other Study IDs: UniversidadeNL_30088; 02/SAICT/2017_30088 (Other: Fundação para a Ciência e a Tecnologia)
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Lung Cancer; Malignancy
Keywords: pleural effusion; thoracentesis; transudate; exudates
MeSH Terms: conditions — Lung Neoplasms; Neoplasms; Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Pleural effusion contains cells. We aim to both characterize the proteome of protein fractions of the acellular pleural effusion and the cellular component. DNA is not the target of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thoracentesis: Patients who need removal of excess pleural effusion and assessed for the possibility of lung cancer.
  Interventions: Diagnostic Test: Proteomics analysis of pleural effusion

INTERVENTIONS:
Diagnostic Test: Proteomics analysis of pleural effusion — Pleural effusion removed as part of standard care is fractionized and analyzed by mass spectrometry

SUMMARY:
The excessive accumulation of fluid between the membranes surrounding the lung, a clinical condition commonly referred to as "pleural effusion", is caused by one of three factors: increased production of pleural fluid, decreased ability to reabsorb pleural fluid or a mixture both.

The basis of pleural effusion accumulation may originate from multiple pathologies: from benign and extrapulmonary conditions to intrinsic pleural pathology (inflammatory or neoplastic primary or metastatic) in which the accumulation of fluid in the pleural space is mainly due to changes in the structure of the pleural membrane (loss of integrity and / or infiltration by neoplastic cells).

An example of extrapulmonary conditions is the pleural effusion observed in patients with congestive heart failure in which there is increase in hydrostatic capillary pressure, due to failure of the cardio circulatory pump.

The distinction between benign and malignant causes is currently a diagnostic challenge that usually requires the collection of material (cells immersed in the pleural fluid or even a histological sample).

The first step of this investigation is currently the cytological evaluation of the pleural fluid, that is, the observation of cells, of an initial sample of the pleural fluid. This procedure is associated with an average sensitivity of 62% while a second sample through thoracentesis improves the sensitivity of the diagnosis by 10%. In certain cases, however, it is not possible to diagnose by analyzing the pleural fluid and, as a rule, a more invasive diagnostic method is recommended, such as pleural biopsy (collected by puncture with a "blind" needle, echo guided or computed tomography guided or obtained by means of direct visualization of the pleural cavity through pleuroscopy).

The diagnostic yield of this approach can reach up to 97% (in the case of pleural biopsy obtained by medical thoracoscopy). However, it implies greater morbidity and greater consumption of resources (material and human). The development of a more sensitive and specific and at the same time less invasive diagnostic method for pleural fluid may contribute to a more effective screening of patients, limiting the use of more invasive methods to only patients with a higher risk of malignant pathology.

DETAILED DESCRIPTION:
The excessive accumulation of fluid between the membranes surrounding the lung, a clinical condition commonly referred to as "pleural effusion", is caused by one of three factors: increased production of pleural fluid, decreased ability to reabsorb pleural fluid or a mixture both.

The basis of pleural effusion accumulation may originate from multiple pathologies: from benign and extrapulmonary conditions to intrinsic pleural pathology (inflammatory or neoplastic primary or metastatic) in which the accumulation of fluid in the pleural space is mainly due to changes in the structure of the pleural membrane (loss of integrity and / or infiltration by neoplastic cells).

An example of extrapulmonary conditions is the pleural effusion observed in patients with congestive heart failure in which there is increase in hydrostatic capillary pressure, due to failure of the cardio circulatory pump.

The distinction between benign and malignant causes is currently a diagnostic challenge that usually requires the collection of material (cells immersed in the pleural fluid or even a histological sample).

The first step of this investigation is currently the cytological evaluation of the pleural fluid, that is, the observation of cells, of an initial sample of the pleural fluid. This procedure is associated with an average sensitivity of 62% while a second sample through thoracentesis improves the sensitivity of the diagnosis by 10%. In certain cases, however, it is not possible to diagnose by analyzing the pleural fluid and, as a rule, a more invasive diagnostic method is recommended, such as pleural biopsy (collected by puncture with a "blind" needle, echo guided or computed tomography guided or obtained by means of direct visualization of the pleural cavity through pleuroscopy).

The diagnostic yield of this approach can reach up to 97% (in the case of pleural biopsy obtained by medical thoracoscopy). However, it implies greater morbidity and greater consumption of resources (material and human). The development of a more sensitive and specific and at the same time less invasive diagnostic method for pleural fluid may contribute to a more effective screening of patients, limiting the use of more invasive methods, only for patients with a higher risk of malignant pathology.

Study Objectives:

This project consists of a preclinical study where we will explore new methodologies for clinical evaluation, based on proteomic analysis of the immunological characteristics and the microenvironment of the tumor in the pleural fluid of patients whose diagnosis has not been confirmed. The results obtained will be used in the implementation of an algorithm for the classification of pleural fluid in the following groups: a) low risk or benign; b) high risk or malignant. If the algorithm has good sensitivity and specificity for malignant diagnoses, it may be useful to distinguish patients in to the groups: a) postpone the invasive test and do active imaging surveillance; b) proceed to invasive testing.

Benefit / Risk Assessment:

The collection of the pleural fluid will be carried out by procedures used in standard care and diagnosis of the disease, thus not constituting additional risks to the participants. The results of this investigation do not bring clinical effects directly applicable to the participants involved. However, in the future the results obtained may benefit other users through improved understanding the tumor microenvironment.

Modalities of Recruitment:

Through an interview with the investigating doctor, the participant in this study becomes aware of the terms of the treatment of his personal data in the scope of the research project. In addition, data subjects sign informed consent for participation in the study. The notification includes an explanation of the procedures involved in the investigation and the role of personal data collected in the context of the investigation. In an interview with the investigating doctor and by signing the informed consent for participation in the study, the data subject becomes aware of his right to withdraw from the study and / or to withdraw his informed consent.

The collection of biological samples for the comparative prospective cohort study will be carried out in all collaborative hospitals in this project in a period of two to three years. Based on the variance and statistical power observed in a previous study of the pulmonary fluid exosome proteome, 200 samples were estimated as the minimum number for the classification of biological samples. The analysis of statistical power is based on the variance observed in 10 samples in which approximately 3500 proteins were identified and quantified in pulmonary fluids. The statistical power analysis considers the correction for multiple tests according to the number of proteins identified and quantified.

Data collection specifications:

During the consultation, a clinical interview will be conducted, which will allow the collection of personal data, namely genetic data, data related to health and racial or ethnic origin. An objective exam will also be carried out to assess weight, height, blood pressure and heart rate. Data relating to the results of complementary diagnostic tests will be collected, namely: 1. Chest X-ray (location, extent and characteristics of the pleural effusion); 2. chest ultrasound (location, extent, characterization of the ecostructure - homogeneous / heterogeneous; with / without visible septations); 3. Thoracic Computed Tomography (location, extent, morphological aspect of the pleura - thickness increase, nodules, etc.); 4. Cytological evaluation of the pleural fluid; 5. Serum biochemical study: blood glucose level; assay of total proteins and serum albumin; lactate dehydrogenase level.

The reference diagnostic method will be based on histological evaluation of the tissue. The results of the proteomics analysis obtained in this project will not be taken into account for the final diagnosis of the participants.

Specification of collection and final destination of biological samples:

According to the clinician's decision, pleural fluid will be obtained for diagnosis (through thoracentesis or during the course of pleural biopsy or pleuroscopy). The sample obtained will follow the usual clinical investigation pathway (cytological and / or histopathological evaluation, biochemical evaluation, microbiological evaluation) as registered in each institution. For patients who agree to participate in the study, only an additional sample of pleural fluid will be sent for the study that we propose to carry out. These last samples will be stored at CEDOC.

Text of information to be provided to volunteers:

The study for which we ask for your consent aims to develop a diagnostic method with greater specificity and sensitivity in identifying different pathologies associated with excessive accumulation of pleural fluid (a condition commonly known as pleural effusion). Currently, the cytological evaluation, that is, the observation of cells, of an initial sample of the pleural fluid has an average sensitivity of 62% while a second sampling through thoracentesis (consists of aspiration of the liquid from the pleura through the puncture of the chest wall) improves the sensitivity of the diagnosis by 10%. In certain cases it is not possible to diagnose by analyzing the pleural fluid and as a rule a more invasive diagnostic method is recommended, such as pleural biopsy or pleuroscopy (surgical technique that allows you to directly view the inside of the rib cage) with pleural biopsy (sensitivity 98%). The development of a diagnostic method with greater specificity and sensitivity of the pleural fluid, thus avoiding invasive methods, can improve the efficiency in screening patients with pleural effusion, limiting the invasive study to a selected portion of patients with an effectively higher risk of malignant pathology. Your participation in this study does not involve additional procedures beyond those that your doctor considers necessary for the diagnosis of the disease or prescription of specific drugs for the study in question. The collected samples will be anonymized with a code, that is, it will not be possible for the researchers to match the samples with the personal data of the respective patients. Any of the data collected will be confidential, in accordance with the new General Data Protection Regulation (GDPR) that came into force last May 2018 (Regulation (EU) No. 2016/679).

PATIENT'S INFOMRED CONSENT:

(NAME) _____________________________________________________, I voluntarily agree to take part of the research project entitled "Clinical study in the context of the diagnosis of patients with pleural effusion".

I declare that I was informed about the objectives and methodology of this study, as well as about the conditions of participation, having received oral and written information, which I heard, read and understood.

This document was signed after all doubts were clarified with the investigating physician and after reflecting on this proposal for participation with unlimited time.

The samples and data will be encrypted, to protect my identity. I am free to refuse to donate my samples and, even after I have given my consent, I will be able to withdraw it at any time if that is my wish. My decision will in no way affect the quality of my clinical follow-up nor will it change my rights as a patient of the ________________________________________________________ (hospital unit).

At any time, I can request generic information about the study for which samples are being used. However, I will not be informed of the concrete results obtained in my samples, since these data are not relevant for my clinical follow-up.

I also authorize the use of biological samples and data collected, anonymously and confidentially, in subsequent research projects, provided they are authorized by the appropriate Ethics Committee.

Signature of Participant: ______________________________________

Date: __ / __ / _____

Investigator's Signature: ______________________________________

Date: __ / __ / _____

Ownership and data protection of participants / confidentiality:

The security measures in the protection of personal data that will be implemented include 1. Pseudonymization and encryption of personal data; 2. Ability to restore availability and access to personal data in a timely manner in the event of an incident; 3. Process for testing, assessing and regularly evaluating the effectiveness of technical and organizational measures to ensure the security of data processing.

ELIGIBILITY:
Inclusion Criteria:

1. Candidate for diagnostic thoracentesis.
2. The General Data Protection Regulation (Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016) and the Law on Personal Genetic Information and Health Information (Decree-Law no. 131/2014) is fulfilled.
3. Participation in the Study is completely voluntary.
4. It is possible to drop out of the study at any time without affecting the quality of medical care.
5. The information obtained from this study may originate scientific publications, without jeopardizing the anonymity of the Participants.
6. During the course of the Study, it is possible to ask the investigators questions that you consider convenient.
7. This study does not impose any cost on the participants.

Exclusion Criteria:

Participants with unstable / severe medical illness (per investigator's judgment), coagulopathies and / or bleeding disorders, immunodeficiency syndromes (primary or acquired - including HIV infection), active and untreated HCV infection, HBV and active history of intravenous drug addictions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects evaluated by thoracentesis at Hospital CUF Descobertas and CUF Infante Santo and at the Local Health Unit of Guarda may participate.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
diagnosis of lung cancer by histological examination of surgically-excised nodules | 6 months
  diagnosis of lung cancer by histological examination of surgically-excised nodules

CONTACTS AND LOCATIONS:
Overall Officials: Rune Matthiesen, PhD, Principal Investigator — Computational and Experimental Biology Group NOVA MEDICAL SCHOOL / FACULDADE DE CIÊNCIAS MÉDICASUNIVERSIDADE NOVA DE LISBOARua Câmara Pestana, 6-6A | 1150-082 Lisboa Portugal
Locations (1):
- Hospital CUF Descorbertas, Lisbon, Parque Das Nacoes, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
In case of publication, clinical parameters will be listed as overall summaries rather than for each individual.